CLINICAL TRIAL: NCT05727397
Title: A Randomized, Double-Masked, Multicenter, Two-Arm Study Comparing the Efficacy and Safety of RC28-E 2mg Versus Aflibercept in Subjects With Wet Age-Related Macular Degeneration
Brief Title: Efficacy and Safety of RC28-E Versus Aflibercept
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28C004
Record Dates: First submitted 2023-01-10; First posted 2023-02-14 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-02

CONDITIONS: Wet Age-related Macular Degeneration
MeSH Terms: interventions — RC28-E protein; aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RC28-E (Experimental): RC28-E 2 mg will be initially injected 3 times at 4 week intervals, then each subject will be injected every 12 weeks unless there is disease activity. If disease activity is identified, the subject will be reassigned to receive injections every 8 weeks thereafter, up to study exit.
  Interventions: Drug: RC28-E
- Aflibercept (Active Comparator): Aflibercept 2 mg will be injected 3 times at 4 week intervals, followed by injections every 8 weeks.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: RC28-E — Ophthalmic solution for intravitreal injection administered as a 2.0mg/50 µL dose.
  Arms: RC28-E
Drug: Aflibercept — Ophthalmic solution for intravitreal injection administered as a 2.0mg/50 µL dose.
  Other Names: Eylea
  Arms: Aflibercept

SUMMARY:
This is a randomized, double-masked, multicenter study comparing the the efficacy and safety of RC28-E injection (a chimric decoy receptor trap fusion protein by dual blockage of VEGF and FGF-2) versus aflibercept in patients with wet age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Sign the consent form, willing and able to comply with clinic visits and study-related procedures;
* 50 years of age or older;
* Diagnosed with wAMD;
* Active CNV lesion of any type (ie, predominantly classic, minimally classic, or occult [including polypoidal choroidal vasculopathy and retinal angiomatous proliferation]) that exhibits all of the following characteristics:

  * The CNV or sequela of the CNV affect the foveal;
  * A total lesion size of ≤12 disc areas on FFA;
  * Evidence of CNV leakage on FFA;
  * Intra and/or subretinal fluid confirmed on OCT;
* BCVA of 78-19 letters using the ETDRS protocol;
* Sufficiently clear ocular media and adequate pupillary dilatation to allow acquisition of good-quality retinal images to confirm diagnosis.

Exclusion Criteria:

For the study eye:

* CNV due to causes other than AMD, such as ocular histoplasmosis, trauma, pathological myopia, angioid streaks, choroidal rupture, or uveitis;
* Any history of macular pathology unrelated to AMD affecting vision or contributing to the presence of intraretinal or subretinal fluid;
* Presence at screening of central serous chorioretinopathy;
* Retinal pigment epithelial tear involving the foveola on day 1;
* Fibrosis or atrophy involves the foveola;
* Subretinal haemorrhage involves the foveola;
* Any concurrent intraocular condition (eg, amblyopia, aphakia, retinal detachment, cataract, diabetic retinopathy or maculopathy, or epiretinal membrane with traction) that, in the opinion of the investigator, could either reduce the potential for visual improvement or require medical or surgical intervention during the study;
* Current vitreous hemonhage or history of vitreous hemorrhage in the study eye within 4 weeks prior to baseline;
* Uncontrolled glaucoma;
* Spherical equivalent of refractive error demonstrating ≥8 diopters of myopia;
* Previous treatment with anti-VEGF therapy within the 3 months period prior to baseline;
* Intraocular use of long-acting corticosteroids during the 6 month period prior to baseline; intraocular use of short or medium-acting corticosteroids during the 3 month period prior to baseline; periocular use of corticosteroids during the 1 month period prior to baseline;
* Use of topical ocular corticosteroids for 60 or more consecutive days within the 3 month period prior to baseline;
* Macular laser treatment, PDT, TTT or other surgical intervention for AMD within the 3 month period prior to baseline;
* Any cataract surgery or treatment for complications of cataract surgery with steroids within the 3 month period prior to baseline; YAG laser capsulotomy within 1 month before baseline;
* Aphakia or pseudophakia with absence of posterior capsule, unless it occurred as a result of YAG posterior capsulotomy;
* Intraocular or refractive surgery within the 3 month period prior to baseline;
* Previous penetrating keratoplasty or vitrectomy or panretinal photocoagulation or radiotherapy;

For the fellow eye or both eyes:

* Non-functioning non-study eye;
* Treatment with anti-VEGF therapy within the 7 day period prior to baseline in the nonstudy eye;
* Any history of idiopathic or autoimmune-associated uveitis in either eye;
* Current active ocular inflammation or suspected or active ocular or periocular infection in either eye;

General exclusion criteria:

* Any major illness or major surgical procedure within 1 month before screening;
* Active cancer within the past 12 months except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, and prostate cancer with a Gleason score of <6 and a stable prostate-specific antigen for >12 months;
* Requirement for continuous use of any medications and treatments indicated as prohibited therapy;
* Systemic anti-VEGF therapy within the 3 month period prior to baseline;
* Use of systemic corticosteroids for 30 or more consecutive days within the 3 months prior to baseline, with the exception of low stable doses of corticosteroids (defined as ≤10 mg/day prednisolone or equivalent dose)；
* Systemic treatment for suspected or active systemic infection on baseline;
* COVID-19 infection within the 4 week period prior to screening; Hospitalization required severe COVID-19 infection within the 12 month period prior to screening;
* HBsAg(+) and HBV DNA>ULN;
* HCV antibody(+); HIV antibody(+); active syphilitic patients;
* Uncontrolled blood pressure, defined as systolic blood pressure >180 mmHg and/or diastolic blood pressure >100 mmHg;
* Stroke (cerebral vascular accident) or myocardial infarction within the 6 month period prior to baseline;
* History of other disease, metabolic dysfunction, physical examination finding, or historical or current clinical laboratory finding giving reasonable suspicion of a condition that contraindicates the use of the investigational drug or that might affect interpretation of the results of the study or renders the patient at high risk for treatment complications in the opinion of the investigator;
* Pregnancy or breastfeeding, or intention to become pregnant during the study;
* History of a severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of RC28-E or to aflibercept injections, study-related procedure preparations (including fluorescein), dilating drops, or any of the anaesthetic and anti-microbial drops used by the patient during the study;
* Participation in an investigational trial that involves treatment with any drug or device (with the exception of vitamins and minerals) within the 3 month period prior to baseline.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-11-29 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in BCVA at week 48; | Baseline, week 48
  BCVA=Best-corrected visual acuity; Measurement of visual acuity with Early Treatment Diabetic Retinopathy Study (ETDRS) charts.

SECONDARY OUTCOMES:
Average change in BCVA from baseline over the period week 36 through week 48; | Baseline, weeks 36, 40, 44 and 48.
  For each subject, this endpoint is defined as the average of the changes from Baseline to Weeks 36, 40, 44 and 48.
Proportion of subjects with q12w injection; | Baseline, week 48
  q12w=every 12 weeks
Proportion of subjects with q12w injection at week 48 within the subjects with no q8w injection need at week 16, week 20; | Week 16, 20, 48
  for subjects randomized to RC28-E group only; q12w=every 12 weeks; q8w=every 8 weeks; A disease activity assessment (DAA) was performed at pre-specified visits (Weeks 16, 20, 28, 32, 40, 44) to identify q8w injection need.
Proportion of subjects with gain in BCVA of 15/10/5/0 letters or more from baseline to week 48; | Baseline, week 48
  Proportion of subjects; BCVA=Best-corrected visual acuity;
Mean change in CST from baseline to week 16, week 48; | Baseline, week 16, 48
  CST=Central retinal subfield thickness
Average change in CST from baseline over the period week 36 through week 48; | Baseline, weeks 36, 40, 44 and 48.
  CST=Central retinal subfield thickness
Proportion of subjects with presence of intraretinal fluid/subretinal fluid at week 16, week 48; | Baseline, week 16, 48
  Intraretinal fluid was assessed using SD-OCT and recorded as Present/Absent. Subretinal fluid was assessed using SD-OCT and recorded as Present/Absent. The presence of intraretinal fluid/subretinal fluid is an indicator of underlying disease.
Percentage of subjects with disease activity present at week 16; | Baseline, week 16
  A disease activity assessment (DAA) was performed to identify q8w injection need. 95% confidence interval (CI) for binomial proportions is based on Clopper-Pearson exact method. One eye (study eye) contributed to the analysis. Hypothesis testing not pre-specified.
Change in choroidal neovascularization (CNV) lesion size from baseline to week 12, week 48; | Baseline, week 12, 48
  CNV lesion size (the area of new blood vessels in the choroid layer of the retina) was measured using fundus fluorescein angiography (FFA). A negative change value indicates a reduction in lesion size, whereas a positive change value indicates an increase. An increase in CNV lesion size may indicate progression of the underlying disease. Only one eye (study eye) contributed to the analysis.
Proportion of subjects with q8w treatment need at weeks 16, 20, 28, 32, 40, 44; | Weeks 16, 20, 28, 32, 40, 44
  q8w=every 8 weeks; A disease activity assessment (DAA) was performed at pre-specified visits (Weeks 16, 20, 28, 32, 40, 44) to identify q8w need. This outcome measure was pre-specified for RC28-E arm only.
Incidence and characteristics of ocular and systemic treatment emergent adverse events. | Baseline, week 48
  safety endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided